CLINICAL TRIAL: NCT03172078
Title: Effects of Target-controlled Infusion and Bispectral Index Monitoring in Sedation of Advanced Endoscopic Procedure
Brief Title: Sedation of Advanced Endoscopic Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201612218RINC
Record Dates: First submitted 2017-05-23; First posted 2017-06-01 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2018-08

CONDITIONS: Sedation
Keywords: advanced endoscopic procedure; ERCP; EUS; target-controlled infusion; sedation; propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Target-control infusion without bispectral index monitoring (Active Comparator): Target-control infusion (TCI) with propofol during advanced endoscopic procedure e.g. endoscopic Ultrasound (EUS), endoscopic retrograde cholangiopancreatogram (ERCP)
  Interventions: Procedure: advanced endoscopic procedure
- Target-control infusion with bispectral index monitoring (Active Comparator): Target-control infusion (TCI) with propofol and BIS monitoring during advanced endoscopic procedure e.g. endoscopic Ultrasound (EUS), endoscopic retrograde cholangiopancreatogram (ERCP)
  Interventions: Procedure: advanced endoscopic procedure

INTERVENTIONS:
Procedure: advanced endoscopic procedure — The advanced endoscopic procedure include endoscopic Ultrasound (EUS), endoscopic retrograde cholangiopancreatogram (ERCP), and other upper gastrointestinal endoscopy.

SUMMARY:
To evaluate the impacts of target-control infusion (TCI) and bispectral index (BIS) monitoring during advanced endoscopic procedure.

DETAILED DESCRIPTION:
Anesthesia requirements for advanced endoscopic procedures are approaching those of specialized surgical interventions. Although many other sedative agents are used prior to and during endoscopy, none approach propofol in terms of desirable properties. The risk of propofol sedation for interventional procedures such as endoscopic retrograde cholangiopancreatography (ERCP), endoscopic ultrasound (EUS), and therapeutic endoscopy are among the highest for any sedated endoscopic procedure. The reasons are many: the intensity of stimulation encountered during these procedures is similar to many minor surgeries; the airway management is complex and requires constant attention; the incidence of hypoxemia is high, and the time available for recognition and management is limited. In order to reap the benefits of advanced endoscopic procedures, anesthesiologists must rise to the challenge. This requires a dedicated anesthetic team practicing safe, efficient, and effective sedation techniques for advanced endoscopic procedures. Ongoing research into novel infusion methods can add safety to the existing sedation techniques and address some of the concerns related to sedative quality. This is a randomized controlled and prospective study. To evaluate the benefits when we use target-controlled infusion of propofol (TCI) with/without bispectral index monitoring in patients undergoing advanced endoscopic procedure. The primary outcome is the total amount of propofol. The secondary outcomes are patients' and endoscopists' satisfaction, sedative-related adverse events, recovery time.

ELIGIBILITY:
Inclusion Criteria:

* patients undergo advanced endoscopic procedure

Exclusion Criteria:

* age less than 20 years, pregnant and lactating women, American Society of Anesthesiologists (ASA) class V, allergy to propofol, benzodiazepine, or opioid, and a requirement for general anesthesia

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-06-05 (Actual); Primary Completion 2018-08-22 (Actual); Study Completion 2018-08-22 (Actual)

PRIMARY OUTCOMES:
propofol dose | during the endoscopic procedure
  Total amount of propofol during the procedure

SECONDARY OUTCOMES:
sedation-related adverse events | during the endoscopic procedure
  hypotension, hypoxemia
Quality of sedation | 2 days
  The satisfaction of the endoscopist with the sedation is evaluated by a case-by-case questionnaire. Four classes of response: excellent, good, acceptable and poor, were defined for the overall evaluation with the safety of endoscopy procedure, patient cooperation and fluency of the procedure in the opinion of the endoscopist. Patients' satisfaction includes their immediate evaluation of side effects such as post procedure dizziness, nausea/vomiting, or pain recall evaluation in the recovery room. Telephone interviews are performed to ascertain the patients' overall satisfaction evaluation and of the procedure with four classes of responses: excellent, good, acceptable and poor.
Recovery: open eye, conscious clear, discharge time | within 2 hrs
  Recovery data include time from end of endoscopy until eye opening on command and time from end of endoscopy until leaving the recovery room based on Aldrete score ≧ 9.

CONTACTS AND LOCATIONS:
Overall Officials: LIN, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No